CLINICAL TRIAL: NCT04316416
Title: Evaluation of The Postoperative Analgesic Effectivity of Erector Spina Plane Block With Different Injection Levels on Patients Undergoing Laparoscopic Cholecystectomy Surgery : A Randomised Controled Study
Brief Title: Evaluation of Effectivity of Erector Spina Plane Block With Different Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, Attending Anesthesiologist, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREH18
Record Dates: First submitted 2020-03-08; First posted 2020-03-20 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; erector spinae plane blok; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- T7 Bilateral ESP block (Active Comparator): Ultrasound-guided bilateral Erector spinae plane block will performe at end of the surgery with 40 ml of a bupivacaine/lidocaine mixture by imaging T7 (7th thoracal vertebrae ) transverse process accompanied by ultrasound. Postoperative routine analgesic protocol planned (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block). Standard pain follow-up and monitorization will be performed.
  Interventions: Procedure: T7 Level Erector Spinae Plane Block
- T9 bilateral ESP block (Active Comparator): Ultrasound-guided bilateral Erector spinae plane block will performe at end of the surgery with 40 ml of a bupivacaine/lidocaine mixture by imaging transverse process T9 (9th thoracal vertebrae) by ultrasound. Postoperative routine analgesic protocol planned (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block). Standard pain follow-up and monitorization will be performed.
  Interventions: Procedure: T9 Level Erector Spinae Plane Block
- Control group (Placebo Comparator): Postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard pain follow-up and monitorization will be performed. No block will be performed in this group.
  Interventions: Drug: control group

INTERVENTIONS:
Procedure: T7 Level Erector Spinae Plane Block — ESP block is planned after the completion of surgery and before the extubation. Its application will be planned from the T7 level bilaterally when the patients are turned to the right lateral position. A linear ultrasound probe will be placed in the longitudinal parasagittal orientation 3 cm to lateral of T7 spinous process.
  After imaging of erector spina musceles and transvers process of 7 th trorocal vertebrae, an ultrasound-guided local anaesthetic mixture ( 0.5% bupivacaine 15 cc + 2% lidocaine 5 cc) will be applied to the region between spinae muscles and transverse process using a needle of 22 gauge & 8cm directed from cranial to caudal.
  After application of the same procedure to the other side, the patients will be woken-up and patient-controlled analgesia consisting of intravenous morphine will be planned for all of them.
  Additionally, at postoperative 1.,4.,8.,12.,24. hours, NRS scales and morphine consumption will be recorded.
  Arms: T7 Bilateral ESP block
Procedure: T9 Level Erector Spinae Plane Block — ESP block is planned after the completion of surgery and before the extubation. Its application will be planned from the T9 level bilaterally when the patients are turned to the right lateral position. A linear ultrasound probe will be placed in the longitudinal parasagittal orientation 3 cm to lateral of T9 spinous process.
  After imaging of erector spina musceles and transvers process of 9 th trorocal vertebrae, an ultrasound-guided local anaesthetic mixture ( 0.5% bupivacaine 15 cc + 2% lidocaine 5 cc) will be applied to the region between spinae muscles and transverse process using a needle of 22 gauge & 8cm directed from cranial to caudal.
  After application of the same procedure to the other side, the patients will be woken-up and patient-controlled analgesia consisting of intravenous morphine will be planned for all of them.
  Additionally, at postoperative 1.,4.,8.,12.,24. hours, NRS scales and morphine consumption will be recorded.
  Arms: T9 bilateral ESP block
Drug: control group — 24 hours morphine consumption will be recorded using the patient controlled analgesia device with intravenous morphine.
  Arms: Control group

SUMMARY:
In last years, erector spinae plane block is widely used in abdominal and thoracic surgeries. Laparoscopic cholecystectomy is one of the most commonly performed surgical operations. In this study, the investigators will evaluate the effectiveness of erector spina plan block with different injection levels for postoperative analgesia on patients undergoing laparoscopic cholecystectomy surgery.

DETAILED DESCRIPTION:
Three groups were planned for this study.Randomization was planned with the closed envelope method. İn the first group, the ESP(erector spinae plane) block procedure will be applied from the T7 level bilaterally and in the second group it will be applied from the T9 level bilaterally. ESP block procedure will not be applied in the third group and this group will be considered as the control group. A comparison of NRS (Numeric Rating Scale) and morphine consumption will be planned for all groups of patients at 1-th, 4-th, 8-th.,12-th and,24-th postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 Elective cholecystectomy surgery
* 18-65 years old patients

Exclusion Criteria:

* ASA 3-4 patients
* Patient refusal
* several lung and heart disease
* Contraindications to regional anesthesia
* BMİ > 35 patients
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Severe kidney or liver disease
* Patient with psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Postoperative pain change | up to 24 hours
  It was planned to check the change in the NRS scores of patients at 1.,4.,8.,12.,24 hours for evaluation of efficacy level and effect time of ESP block procedure from different levels.
  A NRS involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain.
Postoperative morphine consumption change | up to 24 hours
  It was planned to check the change in the morphine consumption of patients at 1.,4.,8.,12.,24 hours for evaluation of efficacy level and effect time of ESP block procedure from different levels.

SECONDARY OUTCOMES:
side effects | up to 24 hours
  Rate of side-effect occurrences (such as rate of vomiting,nausea,shoulder pain) between groups will be compared.
number of blocked dermatome sites | up to 24 hours
  number of blocked dermatome sites will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: SERPİL SEHİRLİOGLU, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital; AYFER KAYA GOK, MD, Study Chair — Gaziosmanpasa Research and Education Hospital; UMRAN YAMAN, MD, Study Chair — Gaziosmanpasa Research and Education Hospital; AYGEN U TURKMEN, MD, Study Chair — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altiparmak B, Toker MK, Uysal AI, Kuscu Y, Demirbilek SG. [Efficacy of ultrasound-guided erector spinae plane block for analgesia after laparoscopic cholecystectomy: a randomized controlled trial]. Braz J Anesthesiol. 2019 Nov-Dec;69(6):561-568. doi: 10.1016/j.bjan.2019.09.001. Epub 2019 Dec 9. PMID 31822353